CLINICAL TRIAL: NCT00979784
Title: The Better Weight-Better Sleep Study: A Pilot Intervention in Primary Care
Brief Title: Better Weight-Better Sleep (BWBS) Trial
Acronym: BWBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Summa Health System (Other)
Collaborators: Northeastern Ohio Universities College of Medicine (Other); Ross Products (Industry)
Responsible Party: Principal Investigator, Everett Logue, Principal Investigator, Summa Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SUMMA-FMRC01
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Overweight; Obesity
Keywords: obesity; primary care
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Behavioral: Better Weight
- 2 (Experimental)
  Interventions: Behavioral: Better Weight & Better Sleep

INTERVENTIONS:
Behavioral: Better Weight — Standard cognitive behavioral treatment focused on dietary & exercise behavior
  Arms: 1
Behavioral: Better Weight & Better Sleep — Standard CBT to support dietary and exercise change plus sleep hygiene and sleep focused CBT
  Arms: 2

SUMMARY:
The hypothesis of this study is that overweight and obese patients exposed to sleep focused counseling and standard dietary and exercise counseling will have better outcomes than similar patients exposed to standard dietary and exercise counseling only.

DETAILED DESCRIPTION:
Objective: To explore the feasibility of integrating sleep management interventions with dietary and exercise interventions for obesity in a 12-week randomized trial. Methods: We randomized 49 overweight or obese adult patients either to a better weight (BW) cognitive behavioral intervention, or to a combination of the BW intervention and a better sleep intervention, better weight-better sleep (BWBS). Results: The BWBS group lost weight faster (P=.04), and coping self-efficacy accelerated (P=.01). Conclusions: These preliminary results merit replication in a larger primary care-based trial with a longer continuous intervention and followup period. Key words: obesity, sleep, weight loss, primary care, health behavior E Logue et al. Am J Health Behav. 2012;36(3):319-334 DOI: http://dx.doi.org/10.5993/AJHB.36.3.4

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 to 39.9
* ages 18 to 84
* PCP permission
* patient in Family Medicine Center with an encounter in the last six months

Exclusion Criteria:

* various obesity and sleep related disorders

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
percent baseline weight lost | 16 weeks

SECONDARY OUTCOMES:
feasibility, variance-covariance estimates | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Family Medicine Center, Summa Health System, Akron, Ohio, United States